CLINICAL TRIAL: NCT02951897
Title: Application of Detecting Circulating Tumor Cells in the Accurate Diagnosis and Treatment of Early Stage Lung Adenocarcinoma
Brief Title: Application of Detecting Circulating Tumor Cells in the Accurate Treatment of Early Stage Lung Adenocarcinoma
Acronym: CTCs detection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Deng Bo, MD, Principal Investigator, Third Military Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMMU-DP-2016-4-25
Record Dates: First submitted 2016-10-25; First posted 2016-11-01 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-10

CONDITIONS: Lung Adenocarcinoma, Stage I; Diagnoses Diseases; Circulating Tumor Cells; Treatment
Keywords: circulating tumor cells; lung adenocarcinoma; treatment; early diagnosis
MeSH Terms: conditions — Adenocarcinoma of Lung; Neoplastic Cells, Circulating; Disease | interventions — Anterior Temporal Lobectomy; Lymph Node Excision

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- IA-CTC-High-enhance (Active Comparator): IA lung adenocarcinoma cases with high abundant CTCs prior to operation will undergo lobectomy&lymphadenectomy plus adjuvant chemotherapy. Postoperative CTC monitoring will be conducted.
  Interventions: Procedure: lobectomy; Drug: chemotherapy（pemetrexed+CISPLATIN）; Procedure: Lymphadenectomy; Other: CanPatrolTM to detect CTCs
- IA-CTC-High-controls (Placebo Comparator): IA lung adenocarcinoma cases with high abundant CTCs prior to operation will only undergo lobectomy&lymphadenectomy. Postoperative CTC monitoring will be conducted.
  Interventions: Procedure: lobectomy; Procedure: Lymphadenectomy; Other: CanPatrolTM to detect CTCs
- IA-CTC-low-controls (Placebo Comparator): IA lung adenocarcinoma cases with low abundant CTCs prior to operation will only undergo segmentectomy. Postoperative CTC monitoring will be conducted.
  Interventions: Procedure: segmentecomy; Other: CanPatrolTM to detect CTCs
- IB-CTC-High-enhance (Active Comparator): IB lung adenocarcinoma cases with high abundant CTCs prior to operation will undergo lobectomy&lymphadenectomy plus adjuvant chemotherapy. Postoperative CTC monitoring will be conducted.
  Interventions: Procedure: lobectomy; Drug: chemotherapy（pemetrexed+CISPLATIN）; Procedure: Lymphadenectomy; Other: CanPatrolTM to detect CTCs
- IB-CTC-High-controls (Placebo Comparator): IB lung adenocarcinoma cases with high abundant CTCs prior to operation will undergo lobectomy&lymphadenectomy. Postoperative CTC monitoring will be conducted.
  Interventions: Procedure: lobectomy; Procedure: Lymphadenectomy; Other: CanPatrolTM to detect CTCs
- IB-CTC-low-controls (Placebo Comparator): IB lung adenocarcinoma cases with low abundant CTCs prior to operation will undergo lobectomy&lymphadenectomy. Postoperative CTC monitoring will be conducted.
  Interventions: Procedure: lobectomy; Procedure: Lymphadenectomy; Other: CanPatrolTM to detect CTCs

INTERVENTIONS:
Procedure: lobectomy
  Arms: IA-CTC-High-controls; IA-CTC-High-enhance; IB-CTC-High-controls; IB-CTC-High-enhance; IB-CTC-low-controls
Procedure: segmentecomy
  Arms: IA-CTC-low-controls
Drug: chemotherapy（pemetrexed+CISPLATIN）
  Arms: IA-CTC-High-enhance; IB-CTC-High-enhance
Procedure: Lymphadenectomy — Lymphadenectomy or lymph node dissection is the surgical removal of one or more groups of lymph nodes. It is almost always performed as part of the surgical management of cancer. In a regional lymph node dissection, some of the lymph nodes in the tumor area are removed; in a radical lymph node dissection, most or all of the lymph nodes in the tumor area are removed.
  Arms: IA-CTC-High-controls; IA-CTC-High-enhance; IB-CTC-High-controls; IB-CTC-High-enhance; IB-CTC-low-controls
Other: CanPatrolTM to detect CTCs — CanPatrol TM was used to detect CTCs, which is a newly established technology to detect CTCs, containing the following steps: (1) To remove erythrocytes by red blood cell lysis and deplete CD45+ leukocytes in 10ml blood sample using a magnetic bead separation method; (2) To enrich CTCs by 8-μm-diameter-pore calibrated membrane filters; and (3) To identify and characterize CTCs by using RNA-in situ hybridization (ISH), based on the branched DNA (bDNA) signal amplification technology, to detect EMT markers, e.g., cytokeratins(CK) 8, 18 and 19, epithelial cell adhesion molecule (EpCAM), vimentin and twist. The details of classification of CTCs by using CanPatrol TM was depicted in the recently published protocol. Finally, the CTCs were clustered into three subtypes, as per the EMT markers, i.e., epithelial (E-) CTCs, mesenchymal (M-) CTCs and epithelial- mesenchymal (E&M-) CTCs.

SUMMARY:
In 2015-2016, 224,390 cases were newly diagnosed with lung cancer in USA. Of all the cases, 83% are non-small cell lung cancer (NSCLC). Currently, the 5-year survival rate of NSCLC patients is 21%, and more than 25% of early stage NSCLC patients, who have undergone surgical treatment, will have a relapse or progression.

Circulating tumor cells (CTCs), which shed from the primary tumor into the vasculature or lymphatics, can be regarded as a new prognostic factors of metastatic process. Thus far, CTCs-detection technologies can be divided into epithelial cell adhesion molecule (EpCAM)-based detection methods, e.g., the widely used CellSearch® and Adnatest®,and EpCAM-independent detection methods, e.g., ISET® and ScreenCell®. Herein, the investigators used a newly established approach, i.e., CanPatrolTM to detect CTCs in early stage lung Adenocarcinoma cases.

The investigator aim to explore whether CTCs detection prior to surgery can be contributive to the early diagnosis, or may help to predict the prognosis and guide the treatment strategy of early stage lung Adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* stage I lung adenocarcinoma

Exclusion Criteria:

* cases with any new adjuvant treatment prior to surgery

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-04; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | From date of diagnosis until the date of first documented progression or date of cancer related death , whichever came first, assessed up to 60 months

CONTACTS AND LOCATIONS:
Locations (1):
- Daping hospital, Chongqing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hofman V, Bonnetaud C, Ilie MI, Vielh P, Vignaud JM, Flejou JF, Lantuejoul S, Piaton E, Mourad N, Butori C, Selva E, Poudenx M, Sibon S, Kelhef S, Venissac N, Jais JP, Mouroux J, Molina TJ, Hofman P. Preoperative circulating tumor cell detection using the isolation by size of epithelial tumor cell method for patients with lung cancer is a new prognostic biomarker. Clin Cancer Res. 2011 Feb 15;17(4):827-35. doi: 10.1158/1078-0432.CCR-10-0445. Epub 2010 Nov 23. PMID 21098695
- [Background] Bayarri-Lara C, Ortega FG, Cueto Ladron de Guevara A, Puche JL, Ruiz Zafra J, de Miguel-Perez D, Ramos AS, Giraldo-Ospina CF, Navajas Gomez JA, Delgado-Rodriguez M, Lorente JA, Serrano MJ. Circulating Tumor Cells Identify Early Recurrence in Patients with Non-Small Cell Lung Cancer Undergoing Radical Resection. PLoS One. 2016 Feb 25;11(2):e0148659. doi: 10.1371/journal.pone.0148659. eCollection 2016. PMID 26913536
- [Background] Sawabata N, Okumura M, Utsumi T, Inoue M, Shiono H, Minami M, Nishida T, Sawa Y. Circulating tumor cells in peripheral blood caused by surgical manipulation of non-small-cell lung cancer: pilot study using an immunocytology method. Gen Thorac Cardiovasc Surg. 2007 May;55(5):189-92. doi: 10.1007/s11748-007-0101-2. PMID 17554991
- [Background] Hofman V, Ilie MI, Long E, Selva E, Bonnetaud C, Molina T, Venissac N, Mouroux J, Vielh P, Hofman P. Detection of circulating tumor cells as a prognostic factor in patients undergoing radical surgery for non-small-cell lung carcinoma: comparison of the efficacy of the CellSearch Assay and the isolation by size of epithelial tumor cell method. Int J Cancer. 2011 Oct 1;129(7):1651-60. doi: 10.1002/ijc.25819. Epub 2011 Mar 11. PMID 21128227
- [Background] Liu L, Liao GQ, He P, Zhu H, Liu PH, Qu YM, Song XM, Xu QW, Gao Q, Zhang Y, Chen WF, Yin YH. Detection of circulating cancer cells in lung cancer patients with a panel of marker genes. Biochem Biophys Res Commun. 2008 Aug 8;372(4):756-60. doi: 10.1016/j.bbrc.2008.05.101. Epub 2008 Jun 2. PMID 18514066
- [Background] Yamashita JI, Kurusu Y, Fujino N, Saisyoji T, Ogawa M. Detection of circulating tumor cells in patients with non-small cell lung cancer undergoing lobectomy by video-assisted thoracic surgery: a potential hazard for intraoperative hematogenous tumor cell dissemination. J Thorac Cardiovasc Surg. 2000 May;119(5):899-905. doi: 10.1016/S0022-5223(00)70084-5. PMID 10788810
- [Background] Nair VS, Keu KV, Luttgen MS, Kolatkar A, Vasanawala M, Kuschner W, Bethel K, Iagaru AH, Hoh C, Shrager JB, Loo BW Jr, Bazhenova L, Nieva J, Gambhir SS, Kuhn P. An observational study of circulating tumor cells and (18)F-FDG PET uptake in patients with treatment-naive non-small cell lung cancer. PLoS One. 2013 Jul 5;8(7):e67733. doi: 10.1371/journal.pone.0067733. Print 2013. PMID 23861795
- [Background] Yoon SO, Kim YT, Jung KC, Jeon YK, Kim BH, Kim CW. TTF-1 mRNA-positive circulating tumor cells in the peripheral blood predict poor prognosis in surgically resected non-small cell lung cancer patients. Lung Cancer. 2011 Feb;71(2):209-16. doi: 10.1016/j.lungcan.2010.04.017. Epub 2010 May 14. PMID 20471712
- [Background] Chen X, Wang X, He H, Liu Z, Hu JF, Li W. Combination of circulating tumor cells with serum carcinoembryonic antigen enhances clinical prediction of non-small cell lung cancer. PLoS One. 2015 May 21;10(5):e0126276. doi: 10.1371/journal.pone.0126276. eCollection 2015. PMID 25996878
- [Background] Yie SM, Lou B, Ye SR, He X, Cao M, Xie K, Ye NY, Lin R, Wu SM, Xiao HB, Gao E. Clinical significance of detecting survivin-expressing circulating cancer cells in patients with non-small cell lung cancer. Lung Cancer. 2009 Feb;63(2):284-90. doi: 10.1016/j.lungcan.2008.05.024. Epub 2008 Jul 7. PMID 18606477
- [Background] Funaki S, Sawabata N, Nakagiri T, Shintani Y, Inoue M, Kadota Y, Minami M, Okumura M. Novel approach for detection of isolated tumor cells in pulmonary vein using negative selection method: morphological classification and clinical implications. Eur J Cardiothorac Surg. 2011 Aug;40(2):322-7. doi: 10.1016/j.ejcts.2010.11.029. Epub 2011 Jan 7. PMID 21215651
- [Background] Yin J, Wang Y, Yin H, Chen W, Jin G, Ma H, Dai J, Chen J, Jiang Y, Wang H, Liu Z, Hu Z, Shen H. Circulating Tumor Cells Enriched by the Depletion of Leukocytes with Bi-Antibodies in Non-Small Cell Lung Cancer: Potential Clinical Application. PLoS One. 2015 Aug 28;10(8):e0137076. doi: 10.1371/journal.pone.0137076. eCollection 2015. PMID 26317979